CLINICAL TRIAL: NCT01931709
Title: Quantitative Dynamic PET and MRI and Breast Cancer Therapy
Brief Title: FDG PET and DCE-MRI in Predicting Response to Treatment in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to end of funding
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Specht, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7587; NCI-2013-01668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7587 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P50CA138293 (NIH); RG1712020 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Male Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Fluorodeoxyglucose F18; Positron-Emission Tomography; Tomography, Emission-Computed; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (FDG PET and DCE-MRI) (Experimental): Patients undergo FDG PET and DCE-MRI 1-2 weeks prior to chemotherapy initiation, between 1-12 weeks after initiation of the first course of chemotherapy, and after the completion of chemotherapy (within 4 weeks prior to surgery).
  Interventions: Radiation: fludeoxyglucose F 18; Device: positron emission tomography; Device: dynamic contrast-enhanced magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo FDG PET
  Other Names: 18FDG; FDG
Device: positron emission tomography — Undergo FDG PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Device: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies fludeoxyglucose F 18 (FDG) positron emission tomography (PET) and dynamic contrast-enhanced (DCE)-magnetic resonance imaging (MRI) in predicting response to treatment in patients with breast cancer. Comparing results of diagnostic procedures done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether detailed kinetic analysis of FDG PET and magnetic resonance (MR) imaging studies for measures of tumor metabolism and blood perfusion can predict response and outcome for breast cancer patients undergoing neo-adjuvant therapy.

II. To compare the in vivo tumor biology associated with responsive and resistant tumors as measured by kinetic changes in FDG PET and MR imaging parameters to tumor subtypes analyzed from assay of pre-therapy biopsy and post-therapy surgical tissue.

OUTLINE:

Patients undergo FDG PET and DCE-MRI 1-2 weeks before prior to chemotherapy initiation, between 1-12 weeks after initiation of the first course of chemotherapy, and after the completion of chemotherapy (within 4 weeks prior to surgery).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer, determined to be a candidate for primary systemic (neoadjuvant) therapy and for surgical resection of residual primary tumor following completion of neoadjuvant therapy
* Primary tumor 2.0 cm or greater, and/or clinical evidence of axillary disease (palpable N1 or N2 or biopsy proven)
* No obvious contraindications for primary chemotherapy
* Able to lie still for PET and MRI scanning
* Able to understand and willing to sign a written informed consent document and a Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines

Exclusion Criteria:

* Serious systemic illness other than breast cancer
* Contraindication to MRI or history of adverse reaction to gadolinium
* Evidence of distant disease outside of regional lymph nodes
* Pregnant
* Poorly controlled diabetes mellitus (fasting blood glucose > 200)
* Prior systemic cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Specht, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Kazerouni AS, Peterson LM, Jenkins I, Novakova-Jiresova A, Linden HM, Gralow JR, Hockenbery DM, Mankoff DA, Porter PL, Partridge SC, Specht JM. Multimodal prediction of neoadjuvant treatment outcome by serial FDG PET and MRI in women with locally advanced breast cancer. Breast Cancer Res. 2023 Nov 9;25(1):138. doi: 10.1186/s13058-023-01722-4. PMID 37946201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (FDG PET and DCE-MRI)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (FDG PET and DCE-MRI)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 43 [31 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Clinical stage [Count of Participants; unit: Participants]
  IIA | 9
  IIB | 8
  IIIA | 9
  IIIB | 3
  IIIC | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Favorable Pathologic Response at Surgery
Description: The primary clinical endpoint is dichotomous (yes/no) - Has patient achieved favorable microscopic pathologic response at surgery? This favorable pathologic response is defined as:
  1. No evidence of microscopic invasive tumor at the primary tumor site and in regional axillary lymph nodes = Residual Cancer Burden class 0 (RCB 0)
  2. Minimal invasive residual disease at primary tumor site and/or in regional axillary lymph nodes = Residual Cancer Burden class I (RCB I)
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (FDG PET and DCE-MRI)
Number analyzed (Participants) | 35
Participants | 11

2. Secondary Outcome: Percent Change in PET K1 Between Mid-therapy and Pre-therapy FDG PET Scans and Its Association With Pathologic Response
Description: Percent change in tumor perfusion between pre-therapy and mid-therapy FDG PET scans as represented by the PET measure K1 (parametric) % change: (Mid-Pre)/Pre, compared between groups of patients who did or did not achieve favorable pathologic response.
Time Frame: Baseline to up to 12 weeks (mid-therapy)
Population: Three participants had to be excluded from this analysis:
  1. mid-therapy PET images got lost due to a technical error;
  2. pre-therapy scanning procedure had 40 seconds delayed start, preventing the modeling of parametric outcomes;
  3. pathologic response could not be evaluated due to a metastatic disease progression prior to surgery.
Measure: Median (Full Range); unit: percent change
Groups:
- Patients With Favorable Pathologic Response: Patients undergo FDG PET and DCE-MRI 1-2 weeks prior to neoadjuvant chemotherapy initiation, between 1-12 weeks after initiation of the first course of chemotherapy, and after the completion of chemotherapy (within 4 weeks prior to surgery).
  Pathologic response at surgery rated as residual cancer burden (RCB) class 0 / I (complete pathologic response or minimal residual disease).
- Patients Without Favorable Pathologic Response: Patients undergo FDG PET and DCE-MRI 1-2 weeks prior to neoadjuvant chemotherapy initiation, between 1-12 weeks after initiation of the first course of chemotherapy, and after the completion of chemotherapy (within 4 weeks prior to surgery).
  Pathologic response at surgery rated as residual cancer burden (RCB) class II /III (moderate to extensive residual disease).
Arm/Group | Patients With Favorable Pathologic Response | Patients Without Favorable Pathologic Response
Number analyzed (Participants) | 10 | 22
percent change | -71.2 [-87.8 to -6.6] | -55.8 [-87.3 to 1035.2]

3. Secondary Outcome: Percent Change in Tumor Metabolism / Perfusion Ratio (MRFDG/K1) Between Mid-therapy and Pre-therapy FDG PET Scans and Its Association With Pathologic Response
Description: Percent change in tumor metabolism / perfusion ratio between pre-therapy and mid-therapy FDG PET scans as represented by the PET measure MRFDG/K1 (parametric) % change: (Mid-Pre)/Pre, compared between groups of patients who did or did not achieve favorable pathologic response.
Time Frame: Baseline to up to 12 weeks (mid-therapy)
Population: as for outcome 2
Measure: Median (Full Range); unit: percent change
Arm/Group | Patients With Favorable Pathologic Response | Patients Without Favorable Pathologic Response
Number analyzed (Participants) | 10 | 22
percent change | -45.0 [-98.1 to 289.2] | -68.5 [-99.2 to 21.9]

4. Secondary Outcome: Time From Surgery to Breast Cancer Recurrence
Description: Mean (range)
Time Frame: The time from surgery to breast cancer recurrence. If recurrence does not occur during follow-up, the endpoint will be censored at the time of last documented disease-free status.
Population: At the time of final analysis, 7 of the 35 patients (20%) had recurrence.
Measure: Mean (Full Range); unit: years- recurrence free
Groups:
- Patients That Received FDG PET and DCE-MRI: Patients were followed for recurrence-free survival and assessed up to 7.5 years.
Arm/Group | Patients That Received FDG PET and DCE-MRI
Number analyzed (Participants) | 7
years- recurrence free | 2.9 [0.4 to 7.5]

5. Secondary Outcome: Time of Surgery to Overall Survival
Description: Mean (range)
Time Frame: Overall survival from time of surgery. If death does not occur during follow-up, the endpoint will be censored at the date of last contact when the patient was verified as alive.
Population: At the time of final analysis, 4 of the 35 patients (11%) had died.
Measure: Mean (Full Range); unit: years- overall survival
Groups:
- Patients That Received FDG PET and DCE-MRI: Patients followed for overall survival and assessed up to 7.5 years
Arm/Group | Patients That Received FDG PET and DCE-MRI
Number analyzed (Participants) | 4
years- overall survival | 3.1 [1.2 to 7.5]

6. Secondary Outcome: Percent Change in DCE-MRI Peak Percent Enhancement (Peak PE) Between Mid-therapy and Pre-therapy Breast MRI Scans and Its Association With Pathologic Response
Description: Percent change in tumor enhancement between pre-therapy and mid-therapy DCE-MRI scans as represented by the MRI measure Peak PE % change: (Mid-Pre)/Pre, compared between groups of patients who did or did not achieve favorable pathologic response.
Time Frame: Baseline to up to 12 weeks (mid-therapy)
Population: One participant had to be excluded from this analysis:
  [1] pathologic response could not be evaluated due to a metastatic disease progression prior to surgery.
Measure: Median (Full Range); unit: percent change
Arm/Group | Patients With Favorable Pathologic Response | Patients Without Favorable Pathologic Response
Number analyzed (Participants) | 11 | 23
percent change | -31 [-49 to -5] | -14 [-63 to 9]

ADVERSE EVENTS:
Arm/Group | Diagnostic (FDG PET and DCE-MRI)
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No